CLINICAL TRIAL: NCT03285880
Title: The Benefits of Naps on Cognitive, Emotional, and Motor Learning in Preschoolers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The pandemic halted the study protocol temporarily. We continued to collect what we could but the study ran out of time/funds.
Sponsor: University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Rebecca Spencer, Associate Professor of Psychological and Brain Sciences, University of Massachusetts, Amherst
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R01HL111695 (NIH)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Within subject comparison of nap and wake conditions
Masking Description: Within-subject; participants/experimenters are aware of conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Declarative memory (Experimental): Napping v. wake effect on a declarative memory task (storybook)
  Interventions: Behavioral: Napping
- Procedural memory (Experimental): Napping v. wake effect on a procedural memory task (motor sequence learning or mirror tracing)
  Interventions: Behavioral: Napping
- Emotional memory (Experimental): Napping v. wake effect on an emotional memory task (emotional faces or storybook)
  Interventions: Behavioral: Napping

INTERVENTIONS:
Behavioral: Napping — Children nap during the nap opportunity

SUMMARY:
The specific objective of the proposed research is to examine whether naps contribute to immediate and delayed benefits on multiple forms of learning in young children (3-5 yrs). By probing recall prior to and following mid-day nap or wake intervals, the overarching hypothesis is that recent memories are actively processed (as opposed to passively protected) by a nap, conferring immediate or delayed (24-hrs) benefits on declarative (Aim 1), procedural (Aim 2), and emotional (Aim 3) memories. In two conditions, children will either be nap-promoted or wake-promoted midday. Subsequently, performance will be reassessed that day as well as the following day.

DETAILED DESCRIPTION:
The proposed research examines whether naps contribute to immediate and delayed benefits on multiple forms of learning in preschool-aged children (3-5 yrs). By probing recall prior to and following mid-day nap or wake intervals, we will examine immediate memory performance and how it is changed by an interval with a nap compared to if that interval was spent awake. There are three arm, separately assessing declarative (using a storybook learning task), procedural (using a mirror tracing task), and emotional (using an emotional storybook task). All children will participate in a nap and wake condition. On the experimental day, children will learn the task, then be nap or wake promoted (within subject, conditions counterbalanced and separated by 1 week). Subsequently, performance will be reassessed that day as well as the following day. Children will wear an actigraph watch for a 16-day interval surrounding the experimental days in order to access habitual sleep patterns (e.g., nap frequency). A subset of children will complete the experimental days in the sleep laboratory. For these children, sleep will be measured using polysomnography, a montage of electroencepholography, electromyography, and electrooculography electrodes.

ELIGIBILITY:
Inclusion Criteria:

* be enrolled in a preschool testing site or available to come into the lab

Exclusion Criteria:

* Diagnosis of any sleep disorder(other than mild parasomnia) past or present
* Current use of psychotropic or sleep-altering medications
* traveling beyond 1 time zone within 1 month of testing
* fever or symptoms of respiratory illness at the time of testing
* physical handicap which interferes with assessments (vision, hearing impairment)
* diagnosed developmental disability

Ages: 33 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 361 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in memory accuracy | 4-5 hours
  Accuracy on the memory task following the nap compared to before the nap relative to the same memory change measured over an interval spent awake

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M Spencer, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurdziel L, Duclos K, Spencer RM. Sleep spindles in midday naps enhance learning in preschool children. Proc Natl Acad Sci U S A. 2013 Oct 22;110(43):17267-72. doi: 10.1073/pnas.1306418110. Epub 2013 Sep 23. PMID 24062429
- [Background] Desrochers PC, Kurdziel LB, Spencer RM. Delayed benefit of naps on motor learning in preschool children. Exp Brain Res. 2016 Mar;234(3):763-72. doi: 10.1007/s00221-015-4506-3. Epub 2015 Dec 8. PMID 26645305
- [Derived] St Laurent CW, Rasmussen CL, Holmes JF, Cremone-Caira A, Kurdziel LBF, Desrochers PC, Spencer RMC. Associations of activity, sedentary, and sleep behaviors with cognitive and social-emotional health in early childhood. J Act Sedentary Sleep Behav. 2023;2(1):7. doi: 10.1186/s44167-023-00016-6. Epub 2023 Apr 3. PMID 38798902
- See also: Lab website — http://www.cognaclab.com